CLINICAL TRIAL: NCT00350493
Title: Three Year Follow up of a Randomised Controlled Trial of an Intervention for Tobacco Dependence Among Those With a Psychotic Illness
Brief Title: Three Year Follow up of a Randomised Controlled Trial (RCT) of an Intervention for Tobacco Dependence Among Those With a Psychotic Illness
Status: Completed | Type: Observational
Sponsor: The University of New South Wales (Other)
Collaborators: Australian Government Department of Health and Ageing (Other Government)
Other Study IDs: 3Yr FollowUp
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Psychotic Disorder; Behavior, Addictive
MeSH Terms: conditions — Psychotic Disorders; Behavior, Addictive

SUMMARY:
This is a three year follow up of a previous study where researchers at UNSW and UNewc asked smokers with serious mental health problems to participate in a 12-month study, to assess whether intervention could assist people experiencing mental illness reduce their tobacco smoking.

DETAILED DESCRIPTION:
Between 2001 and 2003, the School of Public Health and Community Medicine at the University of New South Wales carried out a large study with the Centre for Mental Health Studies at the University of Newcastle. The project asked people with serious mental health problems, who also smoked cigarettes, to participate in a 12-month study, which involved completing several questionnaires/other assessments over that time with a member of the research team. Around half of the participants in this study also received treatment for their smoking from the research team. This treatment involved weekly therapy with one member of the research team, and covered the relationship between smoking and mental illness, teaching people to cope with desires to smoke, how to recognise and avoid high risk situations for smoking, and how to plan alternative ways of coping with those situations where smoking usually occurred. In addition, nicotine patches were also available to assist people who made the decision to reduce their smoking. This study hoped to learn whether this new treatment could assist people experiencing mental illness reduce their tobacco smoking.

After three years, previous participants were invited to participate in another follow-up assessment to check-in with their current situation, their mental health and levels of smoking.

ELIGIBILITY:
Inclusion Criteria:

* Previous participants from the original study

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298
Dates: Start 2005-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Richmond, Professor, Principal Investigator — University of New South Wales; Amanda Baker, Assoc Prof, Principal Investigator — Newcastle University
Locations (2):
- Australia (2):
  - Centre for Mental Health Studies, University of Newcastle, Newcastle, New South Wales
  - School of Public Health and Community Medicine, University of New South Wales, Sydney, New South Wales